CLINICAL TRIAL: NCT02678897
Title: Pain and Medical Abortion - Predicting Factors of Pain and Optimal Pain Management Among Teenaged Women Compared to Adult Women
Brief Title: Pain and Medical Abortion Among Teenaged Women Compared to Adult Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Venla Kemppainen, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS277/03/2015; 2015-003760-36 (EudraCT Number); 2015-005657-12 (EudraCT Number)
Record Dates: First submitted 2015-12-16; First posted 2016-02-10 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Pain
Keywords: Abortion, Drug-Induced; Pain Management
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pain management in early pregnancy MTOP (No Intervention): Patients in early pregnancy (pregnancy weeks <9weeks) undergoing medical termination of pregnancy gets Ibuprofen (tbl 600mg 3 times a day) and Paracetamol (tbl 1000mg 3 times a day).
- Patient controlled analgesia (PCA) (Experimental): Pregnancy weeks 9-20. All patients get baselineanalgesics: Ibuprofein 600mg and Paracetamol 1000mg both x3 a day.
  Patients get pain medication (Oxynorm) via PCA
  Interventions: Drug: Oxynorm via PCA
- Oxynorm on-demand (Active Comparator): Pregnancy weeks 9-20. All patients get baselineanalgesics: Ibuprofein 600mg and Paracetamol 1000mg both x3 a day.
  Patients get extra pain medication (Oxynorm) on-demad from the nurse.
  Interventions: Drug: Oxynorm on-demand

INTERVENTIONS:
Drug: Oxynorm on-demand — We compare different routes of administration (PCA an oral/intramuscular use of oxynorm) in patients undergoing medical termination of pregnancy. Patients are randomized in two groups (for extra pain medication)
  1. If analgesia is inadequate oxycodon (OxyNorm®) (10 mg (less than 80 kg) - 15 mg (over 80 kg) po. In an hour oxycodon 5-10 mg more po if needed. Intramuscular or intravenous administration if needed.
  2. Patient controlled analgesia (PCA pain pump): Oxycodon dose is 3.0 mg (3 ml) and lock-out time 8 min. Maximum four doses in hour. Dose can be lowered or augmented 0,5 mg at time between 2.0-4.0 mg and maximal number of doses can be up to 5.
  Arms: Oxynorm on-demand
Drug: Oxynorm via PCA — We compare different routes of administration (PCA an oral/intramuscular use of oxynorm) in patients undergoing medical termination of pregnancy. Patients are randomized in two groups (for extra pain medication)
  1. If analgesia is inadequate oxycodon (OxyNorm®) (10 mg (less than 80 kg) - 15 mg (over 80 kg) po. In an hour oxycodon 5-10 mg more po if needed. Intramuscular or intravenous administration if needed.
  2. Patient controlled analgesia (PCA pain pump): Oxycodon dose is 3.0 mg (3 ml) and lock-out time 8 min. Maximum four doses in hour. Dose can be lowered or augmented 0,5 mg at time between 2.0-4.0 mg and maximal number of doses can be up to 5.
  Arms: Patient controlled analgesia (PCA)

SUMMARY:
In this two-parted study the need and sufficiency of analgesics and experienced pain is compared between teen-aged and adult women undergoing medical termination of pregnancy (MToP)in early pregnancy (under 9weeks of gestation). During MToP at pregnancy weeks 9-20 on-demand administration of opiates and patient-controlled analgesia (PCA) are compared in randomized clinical trial.

DETAILED DESCRIPTION:
Adequate pain control is crucial in medical abortion. Experience of painful and traumatic abortion can affect patients future plans on pregnancy and childbirth. Study's purpose is to investigate only pain experience and pain management. Otherwise the care of abortion is according to present Finnish national guideline.

Study's goal is to evaluate experienced pain and the need and adequacy of analgesics and to obtain more efficient analgesics during MToP. In addition investigators hope to recognize predicting factors of severe pain.

Study is done in cooperation with Helsinki university and Helsinki university central hospital and is accomplished in Womens hospital and Kätilöopisto hospital in which care of abortions is centralized in HUS area.

Altogether 340 women, who are primigravid, aged between 15-19 or 25-35 years and tolerate used analgesics, are recruited in the study. MToP is done with the combination on mifepristone 200mg and misoprostol 800ug according to Finnish national guidelines. Baseline analgesics are Ibuprofein 600mg ja Paracetamol 1000mg, both three times a day and first dose is taken simultaneously with Misoprostol.

First part is a prospective study in which we compare pain experience and sufficiency of analgesics during MToP in early pregnancy (under 9 weeks of pregnancy). Pain is measured by VAS, which is reported in a diary every time analgesics are needed.

Second part is a controlled randomized study with PCA and on-demand pain management during medical termination of pregnancy with gestational age of 9 to 20 weeks. Every teen-aged woman has two adult controls.

Against severe pain patients get Opiates (oxycodone). In intervention group patients get PCA with Oxycodon dose of 3.0 mg maximal four times in an hour. In control group Oxycodon is administrated on demand po, im or iv depending on the intensity of pain. Pain is measured by VAS from the onset of pain and repeated every 30 minutes until fetal expulsion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who choose medical method of abortion
* First pregnancy
* Age between 15 and 19 years or 25 and 35 years
* Patients volunteer in the study

Exclusion criteria for inquiry part are

* Patient's serious illness
* Known allergy to one of the trial medications
* Abortion is done based on foetal abnormality or threat of patient's own health

Exclusion criteria for intervention part are

* Abortion is done based on foetal abnormality or threat of patient's own health
* Minor patient does not want to inform guardian
* More than one foetus
* Patient's serious illness (ASA-class 3 or 4)
* Massive obesity (BMI >35 kg/m2)
* Known allergy to one of the trial medications
* History of opioid abuse
* Problems of understanding (Inability of use PCA or to understand VAS)
* Active bleeding before intake of first Misoprostol dose
* One of next medications: ketokonatsol, erythromycin, claritromycin, verapamil or diltiazem or medication against HIV (CYP3A4-transmitted interaction with oxycodon)

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 242 (Actual)
Dates: Start 2016-03; Primary Completion 2018-08 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Patients are less painful using patient controlled analgesia (PCA) | During drug-induced abortion, in hospital care (1-2days)
  Measured in visual analog scale (VAS, 0-100mm). VAS is lower.

SECONDARY OUTCOMES:
Patient satisfaction is higher | just after the abortion and 2-3 weeks after in follow-up visit
  Measured in visual analog scale (VAS, 0-100mm), VAS is higher.

OTHER OUTCOMES:
Teen-aged women experience more severe pain than their adult comparators. | during drug-induced abortion
  Measured: Age, visual analogue scale (pain-VAS) is higher during medical abortion.
Patients with history of dysmenorrhea or anxiety experience more severe pain during drug-induced abortion. | During drug-induced abortion
  VAS-scale asked about pain during menstrual bleeding, Anxiety questionnaire (GHQ12, anxiety level is higrher) and Visual analogue scale (VAS) of pain during medical abortion is higher

CONTACTS AND LOCATIONS:
Overall Officials: Oskari Heikinheimo, Professor, Study Director — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Central hospital, Kätilöopistohospital, Helsinki, HUS
  - Helsinki University central hospital, Naistenklinikka, Helsinki, HUS

IPD SHARING:
Plan to Share IPD: No